CLINICAL TRIAL: NCT07274761
Title: A Phase II, Single-arm, Single-center Study of Neoadjuvant Sunvozertinib for Stage II-IIIB Non-small Cell Lung Cancer With EGFR Exon 20 Insertion Mutations.
Brief Title: Neoadjuvant Sunvozertinib in Stage II-IIIB Non-small Cell Lung Cancer Harboring EGFR Exon 20 Insertion Mutation.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-035
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Potentially Resectable EGFR Exon 20 Insertion Non-Small Cell Lung Cancer; Non Small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer stage II-IIIB; Sunvozertinib; EGFR Exon 20 insertion; neoadjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunvozertinib 300 mg orally, once daily (Experimental)
  Interventions: Drug: Sunvozertinib

INTERVENTIONS:
Drug: Sunvozertinib — Participants will receive oral administration of sunvozertinib 300 mg QD, with each treatment cycle defined as 28 days, until meeting any treatment discontinuation criteria.

SUMMARY:
To assess the efficacy and safety of sunvozertinib as neoadjuvant therapy in patients with stage II-IIIB non-small cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) exon 20 insertion mutations (exon20ins).

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient must understand the trial requirements and contents, and provide written informed consent.

  2.Age ≥ 18 years. 3.Histologically or cytologically confirmed non-squamous non-small cell lung cancer (NSCLC). Assessed as resectable Stage II-III disease (per the American Joint Committee on Cancer (AJCC) 8th edition).

  4.Confirmed EGFR exon 20 insertion mutation by a validated test. 5.No evidence of disease progression within the past two weeks prior to signing informed consent and an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

  6.Adequate hematological and organ function, as defined by: 7.Hematological: Absolute Neutrophil Count (ANC) ≥ 1.5 × 10^9/L Platelet count ≥ 100 × 10^9/L Hemoglobin ≥ 9 g/dL

Hepatic:

Total bilirubin ≤ 1.5 × Upper Limit of Normal (ULN); for patients with Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases, total bilirubin ≤ 3 × ULN.

Alanine Aminotransferase (ALT) ≤ 2.5 × ULN and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN in the absence of liver metastases; or ALT and AST ≤ 5 × ULN for patients with liver metastases.

Renal:

Serum creatinine ≤ 1.5 × ULN, AND Calculated or measured creatinine clearance ≥ 60 mL/min (using the Cockcroft-Gault formula).

8.Male patients with female partners of childbearing potential must agree to use a highly effective barrier method of contraception (e.g., condom) during the trial intervention period and for 6 months after the last dose. Male patients must refrain from donating sperm during this same period.

9.Female patients must agree to use contraception from the time of screening until 6 weeks after the last dose, must not be breastfeeding, and must have a negative pregnancy test (serum or urine beta-human chorionic gonadotropin, β-hCG) at screening.

Exclusion Criteria:

* 1.Prior systemic anti-tumor therapy, including chemotherapy, targeted therapy, immunotherapy, and investigational agents from other clinical trials.

  2.History of other malignancies within the past 2 years (except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix).

  3.History of stroke or intracranial hemorrhage within 6 months prior to the first dose.

  4.Severe or uncontrolled systemic diseases/active infection. 5.Any severe or poorly controlled systemic disease, in the investigator's judgment, including but not limited to the following cardiac conditions or abnormalities: QT interval corrected using Fridericia's formula (QTcF) > 470 msec at rest on electrocardiogram (ECG).

Any clinically significant abnormalities in cardiac rhythm, conduction, or morphology at rest on ECG, such as complete left bundle branch block, third-degree atrioventricular block, second-degree atrioventricular block, PR interval > 250 msec.

Any factors that increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death in a first-degree relative under 40 years of age, or any other known condition associated with prolonged QT interval.

Presence of atrial fibrillation (except for drug-induced atrial fibrillation which has resolved after discontinuation of the causative agent).

Myocardial infarction ≤ 6 months prior to the first dose, New York Heart Association (NYHA) Class II or higher congestive heart failure, or poorly controlled arrhythmia despite medical treatment.

6.History of interstitial lung disease (ILD), drug-induced ILD, or any evidence of ILD on imaging at screening.

7.Refractory nausea and vomiting, chronic gastrointestinal diseases, or significant bowel resection that would preclude adequate absorption of Sunvozertinib.

8.Women who are breastfeeding or pregnant. 9.Known hypersensitivity to the active ingredient or any excipients of Sunvozertinib.

10.Patients who, in the judgment of the investigator, are unsuitable for participation in this clinical trial or are unlikely to comply with the study procedures and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 30 months
  ORR is defined according to the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Major pathologic response (MPR) rate | Up to 30 months
Pathological complete response (pCR) rate | Up to 30 months
Event-free suvival (EFS) | Up to 60 months
Overall suvival (OS) | Up to 60 months
R0 resection rate | Up to 30 months
N2 downstaging rate after neoadjuvant treatment | Up to 30 months
Treatment-related adverse event (TRAE) | Up to 30 months
Incidence of treatment discontinuation due to AE/SAE | Up to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.